CLINICAL TRIAL: NCT06760169
Title: Efficacy and Safety of the ELIOS Laser in Combined Cataract and Glaucoma Surgery
Acronym: ELIOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Privé de la Baie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-32-PDB
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma
Keywords: glaucoma; ELIOS laser; micro-invasive surgery; goniotomy
MeSH Terms: conditions — Glaucoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elios (Experimental)
  Interventions: Device: Surgery with ELIOS laser

INTERVENTIONS:
Device: Surgery with ELIOS laser — This surgery involves visualizing the iridocorneal angle before or after cataract surgery, inserting the ELIOS laser probe into the anterior chamber to come into slight contact with the trabecular meshwork, then pressing the foot pedal, the surgeon activates the laser, which creates a microchannel by photoablating the trabecular meshwork and inner wall of Schlemm´s canal (trabeculostomy) ± 210 um in diameter. This gesture is repeated until 10 microchannels are created. The creation of these microchannels enhances the natural outflow of aqueous humor by bypassing the site of major resistance in the system. The usual duration of the ELIOS procedure is typically few minutes). The rest of the surgery does not deviate from standard phacoemulsification.

SUMMARY:
Glaucoma is an irreversible optic neuropathy. It is the second most common cause of blindness worldwide. Glaucoma can be treated with topical medications (eye drops), laser or surgery. Traditional surgery is invasive and has a high complication rate (hypotonia, endophthalmitis, cataracts, etc.). As a result, several types of micro-invasive surgery (MIGS) have been developed to reduce the risks of surgery while maintaining their effectiveness in lowering intraocular pressure (IOP). The ELIOS laser system is the only ophthalmological excimer laser designed for the surgical treatment of glaucoma. The aim of the procedure is to ablate the trabecular meshwork and inner wall of Schlemm´s canal ab interno, with the creation of 10 microchannels of 210 um in the trabeculum using the ELIOS laser with a wavelength of 308 nm, in order to improve trabecular outflow to achieve a reduction in IOP. The ELIOS laser is an example of Microinvasive Glaucoma surgery (MIGS) with published results demonstrating efficacy and safety. The ELIOS laser is already in use in France (AMM / CE mark achieved). Its use as part of a prospective interventional study will enable us to collect data in order to treat patients more effectively and improve the quality of care provided to glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age who agree to take part in the study and have signed an informed consent form
* Visually significant cataract with indication for surgery
* Primary open-angle glaucoma, or secondary open-angle glaucoma (pseudoexfoliative glaucoma or pigmentary glaucoma) with indication for cataract surgery.
* Open iridocorneal angle (Shaffer classification grade 2-4)
* Early to moderate glaucoma (advanced glaucoma, with MD from VFs worse than -12dB, will be excluded)

Exclusion Criteria:

* Presence of severe systemic pathologies 2024-A01891-46_Protocol_V6_21112024_Elios Page 20 / 58
* Pregnant or breastfeeding women
* <18 years of age
* Presence of other ophthalmological pathologies (except cataracts), and exclusion of severe dry eye.
* History of intraocular surgery, trauma, or conjunctival scarring in the quadrant intended for surgery
* Visual acuity worse than "counting fingers".
* Closure of the iridocorneal angle (and angle-closure glaucoma), angle-closure glaucoma secondary to iridocorneal synechiae, neovascular glaucoma or neovascularization of the iris.
* Normal-pressure glaucoma
* Pachymetry < 490 um or > 620 μm
* Glaucomatous visual field with mean deviation worse than ≤-12 dB
* IOP > 35 mmHg
* Autoimmune disorder, especially collagenosis
* Patient under protective supervision
* Patient not covered by a social security scheme

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | day 0, 7 and 30, and month 3, 6 and 12 months after surgery
  This IOP measurement will be carried out using the Goldmann gold standard tonometer, in 2 measurements taken between 8am and 12am, and measured in mmHg

SECONDARY OUTCOMES:
Quality of life | before and after surgery (1, 3, 6 and 12 months)
  A quality of life questionnaire : 25 questions with Likert scales

IPD SHARING:
Plan to Share IPD: No